CLINICAL TRIAL: NCT04166383
Title: Phase II Trial of VB-111 in Combination With Nivolumab in Patients With Metastatic Colorectal Cancer (mCRC).
Brief Title: VB-111 in Combination With Nivolumab in People With Metastatic Colorectal Cancer (mCRC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200022; 20-C-0022
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Cancer With Hepatic Metastases; Colorectal Tumors
Keywords: Nonreplicating adenovirus; Antitumor Immunity; PD-1 inhibition; Immune Checkpoint Inhibition
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Arm 1 (Experimental): Vascular Biogenics (VB)-111 and nivolumab
  Interventions: Biological: Vascular Biogenics (VB)-111; Drug: Nivolumab

INTERVENTIONS:
Biological: Vascular Biogenics (VB)-111 — 1E13 or 0.7E13 VP via intravenous (IV) infusion on Day 1 of cycle 1 and continue every 6 weeks
Drug: Nivolumab — 240 mg of nivolumab via intravenous (IV) infusion on Day 1 of each cycle starting on cycle 2 and continue every 2 weeks
  Other Names: Opdivo

SUMMARY:
Background:

Gastrointestinal cancer is one of the most common cancers worldwide. Researchers think an unmet need exists to understand and improve treatment options. They want to see if a combination of drugs can help people with metastatic colorectal cancer.

Objective:

To see if using a combination of Vascular Biogenics (VB)-111 and nivolumab is safe and will cause colorectal tumors to shrink.

Eligibility:

People ages 18 and older with microsatellite stable colorectal cancer that has spread to the liver

Design:

Participants must consent to sample collection protocol 11C0112.

Participants will be screened with:

Blood tests

Scans

Tumor samples. If these are not available, participants will have a biopsy.

Before they start treatment and with every treatment cycle, participants will have:

Physical exams

Blood tests

Heart tests

Before they start treatment and every 4 cycles, participants will have computed tomography (CT) or magnetic resonance imaging (MRI) scans. For these, they will lie in a machine that takes pictures of the body. For the MRI, a soft padding or coil will be placed around their head.

Participants will have biopsies before they start therapy. They will have them again after 2 6 weeks on study.

On day 1 of 14-day cycles, participants will get one or both study drugs by vein.

After they finish treatment, participants will have monthly visits for 3 months. They will have a physical exam and blood tests.

If participants stop treatment for reasons other than their disease getting worse, they will have scans about every 8 weeks. This will continue until their disease gets worse.

Participants will be contacted by phone or email every 6 months. This will continue for life.

...

DETAILED DESCRIPTION:
Background:

* Immune based approaches in gastrointestinal (GI) cancers have unfortunately- with the notable exception of immune checkpoint inhibition in microsatellite instable (MSI-H) disease and gastric cancer-been largely unsuccessful. The reasons for this are unclear but no doubt relate to the fact that in advanced disease GI cancer appears to be less immunogenic, as evidenced by the lack of infiltrating lymphocytes with advancing T stage as well as an immunosuppressive tumor micro-environment.
* Vascular Biogenics (VB)-111 is an anti-angiogenic agent comprising of a nonreplicating E1 deleted adenovirus type 5 which contains a modified murine preproendothelin (PPE) promoter and Fas-chimera transgene
* VB-111 has been tested and shows promise in glioblastoma, ovarian and thyroid tumors
* Nivolumab is a human monoclonal antibody directed against programmed cell death protein 1 (PD-1).
* The aim of this study is to study the effects of VB-111 in colorectal cancer (CRC) and to evaluate whether the antitumor immunity induced by VB-111 therapy can be enhanced by PD-1 inhibition.

Objectives:

* To determine the safety and tolerability of VB-111 in combination with nivolumab in patients with refractory, metastatic CRC
* To determine Best Overall Response (BOR) (partial response (PR) + complete response (CR)) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) of combined treatment of VB-111 and nivolumab in patients with refractory, metastatic CRC.

Eligibility:

* Histopathological confirmation of colorectal cancer metastatic to the liver
* Patients must have progressed on > 2 lines of standard of care chemotherapy for colorectal cancer or been intolerant of chemotherapy or refused prior chemotherapy.
* Patient's tumors must be documented to be microsatellite stable (MSS).
* Patients must have at least 1 focus of metastatic disease that is amenable to pre-and on-treatment biopsies and be willing to undergo this.
* All patients enrolled will be required to have measurable disease by RECIST v 1.1 criteria.

Design:

* The proposed study is a phase II study of VB-111 in combination with immune checkpoint inhibition (nivolumab) in patients with metastatic CRC
* Treatment will be delivered in cycles consisting of 2 weeks with VB-111 given every 6 weeks and nivolumab given every 2-week until progression or unacceptable toxicity.
* Disease status evaluation will be done every 8 (+/- 1) weeks after the start of study therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histopathological confirmation of colorectal cancer.
* Patients must have radiologically confirmed liver metastasis.
* Patients must:

  * have progressed on > 2 lines of standard of care chemotherapy for colorectal cancer

OR

--been intolerant of standard of care chemotherapy for colorectal cancer

OR

* refused prior standard of care chemotherapy for colorectal cancer.

  * Patients who have a known Kirsten rat sarcoma (KRAS) wild type tumor must have progressed, been intolerant of or refused anti-epidermal growth factor receptor (EGFR) based treatment.
  * Patient's tumors must be documented to be microsatellite stable (MSS).
  * Patients must have at least 1 focus of metastatic disease that is amenable to pre- and on-treatment biopsies and be willing to undergo this. Ideally, the biopsied lesion should not be one of the target measurable lesions, although this can be up to the discretion of the investigator's
  * Patients must have measurable disease by RECIST v 1.1 criteria.
  * Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of nivolumab in combination with Vascular Biogenics (VB)-111 in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-1
  * Adequate hematological function defined by:
* white blood cell (WBC) count greater than or equal to 3x10(9)/L
* absolute neutrophil count (ANC) greater than or equal to 1.5x10(9)/L
* lymphocyte count greater than or equal to 0.5x10(9)/L
* platelet count greater than or equal to 100x10(9)/L
* Hemoglobin (Hgb) greater than or equal to 9 g/ dL (more than 48 hours post-completion of blood transfusion)

  * Prothrombin time (PT) and Partial thromboplastin time (PTT) (seconds) < 1.2 x ULN. Patients who are anticoagulated do not need to meet criteria for PT and PTT
  * International normalized ratio (INR) < 1.2 x ULN. Patients who are anticoagulated do not need to meet criteria for INR.
  * Adequate hepatic function defined by:
* a total bilirubin level less than or equal to 1.5 x ULN,
* an Aspartate transaminase (AST) level less than or equal to 2.5xULN in the absence of hepatic metastasis; or less than or equal to 5 x ULN in the presence of hepatic metastases,
* an Alanine transferase (ALT) level less than or equal to 2.5xULN in the absence of hepatic metastasis; or less than or equal to 5 x ULN in the presence of hepatic metastases

  -Adequate renal function defined by:
* Creatinine OR Measured or calculated creatinine clearance (CrCl) (estimated glomerular filtration rate (eGFR) may also be used in place of CrCl) (A Creatinine clearance (CrCl) or eGFR should be calculated per institutional standard.):

  * < 1.5x institution upper limit of normal OR

greater than or equal to 50 mL/min/1.73 m(2) for participant with creatinine levels greater than or equal to 1.5 X institutional ULN

* The effects of nivolumab and VB-111 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation and up to 5 months (women) and 7 months (men) after the last dose of the nivolumab or 2 months after the last dose of VB-111 whichever is the longer time period. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Troponin level in normal range at the time of enrollment.
* Patient must be able to understand and willing to sign a written informed consent document.
* Weight > 35kg
* Patients must be enrolled in tissue collection protocol 11C0112.

EXCLUSION CRITERIA:

* Patients who have had standard-of-care anti-cancer therapy or therapy with investigational agents (e.g., chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies or other investigation agents), large field radiotherapy, or major surgery within 4 weeks prior to enrollment.
* Patients who have had anti-vascular endothelial growth factor (VEGF) therapy within 4 weeks prior to enrollment.
* Patients currently on a corticosteroid dose greater than physiologic replacement dosing defined as 10 mg of cortisone per day or its equivalent.
* Patients with known brain metastases because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with signs of liver failure, e.g., clinically significant ascites, encephalopathy, or variceal bleeding within 6 months prior to enrollment.
* Prior major liver resection: remnant liver <50% of the initial liver volume. Patients with a biliary stent can be included.
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome or Chronic Inflammatory Demyelinating Polyneuropathy (CIDP), myasthenia gravis; systemic autoimmune disease such as Systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome. Such diseases should be excluded because of the risk of recurrence or exacerbation of disease.

Of note, patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.

* History of idiopathic pulmonary fibrosis (including bronchiolitis obliterans with organizing pneumonia) or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations (within timeframes identified in the bullets below) that would limit compliance with study requirements.
* History of severe or unstable cerebrovascular disease.
* Pulse oximetry < 92% on room air
* Myocardial infarction within 6 months prior to enrollment
* History of myocarditis
* Sustained hypotension (<90/50 mmHg) or uncontrolled hypertension (>160/100 mmHg)
* Stroke within 6 months prior to enrollment.
* Patients with proliferative and/or vascular retinopathy.
* Significant vascular disorders (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to enrollment.
* History of hemoptysis (> 1/2 teaspoon of bright red blood per episode) or active gastrointestinal (GI) bleeding within 6 months prior to enrollment.
* Evidence of a bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to enrollment.
* Human immunodeficiency virus (HIV)-positive patients are excluded because HIV causes complicated immune deficiency and study treatment can possess more risks for these patients.
* Prior autologous or allogenic hematopoietic stem cell transplant.
* Subjects with ascites.
* Patients with unhealed surgical wounds for more than 30 days.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab or VB-111.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years prior to enrollment.
* Pregnant women are excluded from this study because nivolumab and VB-111 potential for teratogenic or abortifacient effects are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab and VB-111, breastfeeding should be discontinued if the mother is treated with nivolumab and/or and VB-111.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-09 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Derived] Coffman-D'Annibale K, Myojin Y, Monge C, Xie C, Hrones DM, Wood BJ, Levy EB, Kleiner D, Figg WD, Steinberg SM, Redd B, Greten TF. VB-111 (ofranergene obadenovec) in combination with nivolumab in patients with microsatellite stable colorectal liver metastases: a single center, single arm, phase II trial. J Immunother Cancer. 2024 Jan 6;12(1):e008079. doi: 10.1136/jitc-2023-008079. PMID 38184304
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0022.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Colorectal Cancers Metastasized to the Liver: Participants with colorectal cancers metastasized to the liver who received Vascular Biogenics (VB)-111 and nivolimab. Second biopsy: Cycle 2 Day 1. VB-111 will be given on Day 1 of cycle 1 and continue every 3 cycles (cycles 4, 7, 10 and so on) at a flat dose of 1x10^13 or 0.7x10^13 viral particles (VP). Nivolumab will be given on day 1 of every cycle starting at cycle 2 at a flat dose of 240 mg. Nivolumab will be administered over approximately 30-60 minutes via intravenous infusion.
  TAC = Treatment Assignment Code
Period: Drug Administration
Arm/Group | Colorectal Cancers Metastasized to the Liver
Started | 14
Completed | 13
Not Completed | 1
Not completed — Prior to treatment (tx), had a medical emergency requiring surgery & was unable to have further tx. | 1
Period: TAC 1 - Second Biopsy Cycle 2 Day 1
Arm/Group | Colorectal Cancers Metastasized to the Liver
Started | 9
Completed | 7
Not Completed | 2
Not completed — Did not complete 2nd biopsy. | 2
Period: TAC 2 - Second Biopsy Cycle 4 Day 1
Arm/Group | Colorectal Cancers Metastasized to the Liver
Started | 5
Completed | 4
Not Completed | 1
Not completed — Did not complete 2nd biopsy. | 1

BASELINE CHARACTERISTICS:
Groups:
- Colorectal Cancers Metastasized to the Liver: Participants with colorectal cancers metastasized to the liver who received Vascular Biogenics (VB)-111 and nivolimab. Second biopsy: Cycle 2 Day 1. VB-111 will be given on Day 1 of cycle 1 and continue every 3 cycles (cycles 4, 7, 10 and so on) at a flat dose of 1x10^13 or 0.7x10^13 viral particles (VP). Nivolumab will be given on day 1 of every cycle starting at cycle 2 at a flat dose of 240 mg. Nivolumab will be administered over approximately 30-60 minutes via intravenous infusion.
Arm/Group | Colorectal Cancers Metastasized to the Liver
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.87 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 1, Grade 2, Grade 3, Grade 4, and/or Grade 5 Adverse Events That Are Possibly, Probably and/or Definitely Related to Drug
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE)v5.0. Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: 90 days after treatment
Population: One participant never treated with study drugs.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 1 Possibly Related; Grade 1 Probably Related; Grade 1 Definitely Related: Grade 1 is mild.
- Grade 2 Possibly Related; Grade 2 Probably Related; Grade 2 Definitely Related: Grade 2 is moderate.
- Grade 3 Possibly Related; Grade 3 Probably Related; Grade 3 Definitely Related: Grade 3 is severe.
- Grade 4 Possibly Related; Grade 4 Probably Related; Grade 4 Definitely Related: Grade 4 is life-threatening.
- Grade 5 Possibly Related; Grade 5 Probably Related; Grade 5 Definitely Related: Grade 5 is death related to adverse event.
Arm/Group | Grade 1 Possibly Related | Grade 1 Probably Related | Grade 1 Definitely Related | Grade 2 Possibly Related | Grade 2 Probably Related | Grade 2 Definitely Related | Grade 3 Possibly Related | Grade 3 Probably Related | Grade 3 Definitely Related | Grade 4 Possibly Related | Grade 4 Probably Related | Grade 4 Definitely Related | Grade 5 Possibly Related | Grade 5 Probably Related | Grade 5 Definitely Related
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13
Participants
  Activated partial thromboplastin time prolonged | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anorexia | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 2 | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fever | 1 | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Flu like symptoms | 0 | 0 | 3 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoxia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mucositis oral | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Other, tachypnea | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sinus tachycardia | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting | 0 | 4 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Best Overall Response (BOR)
Description: Best overall response is defined as the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started) assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions). Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: Follow up visits are planned to be performed at 60 (+/- 14 days) and 90 (+/- 14 days) days after treatment discontinuation to evaluate patient's safety, up to 6 months.
Population: One participant not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Cancers Metastasized to the Liver
Number analyzed (Participants) | 13
Participants
  Complete Response | 0
  Partial Response | 0
  Progressive Disease | 11
  Stable Disease | 2
Statistical Analysis 1: Comparison: Colorectal Cancers Metastasized to the Liver; Test type: Other; p = 0.10, Kaplan-Meier — P≤0.10 (alpha 0.1); power = 90% (beta 0.1)

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival was assessed by the Kaplan-Meier technique with GraphPad Prism 9.3.1 for Windows (GraphPad, San Diego, CA) to calculate these values, and the median PFS will be reported along with 95% confidence interval. PFS is defined as the time between the first day of treatment to the day of disease progression. Disease progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions). Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: The time between the first day of treatment to the day of disease progression, an average of 1.8 months.
Population: One participant never treated with study drugs.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Colorectal Cancers Metastasized to the Liver
Number analyzed (Participants) | 13
Months | 1.8 [0.75 to 2.72]

4. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival was assessed by the Kaplan-Meier technique with GraphPad Prism 9.3.1 for Windows (GraphPad, San Diego, CA) to calculate these values, and the median OS will be reported along with 95% confidence intervals. Overall survival is the time between the first day of treatment to the day of death.
Time Frame: The time between the first day of treatment to the day of death, an average of 6.9 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Colorectal Cancers Metastasized to the Liver
Number analyzed (Participants) | 13
Months | 6.9 [2.64 to 10.74]

5. Secondary Outcome: 6-month Progression-free Survival (PFS)
Description: 6-month progression-free survival was assessed by the Kaplan-Meier technique with GraphPad Prism 9.3.1 for Windows (GraphPad, San Diego, CA) to calculate these values, and the median PFS will be reported along with 95% confidence interval. PFS is defined as the time between the first day of treatment to the day of disease progression. Disease progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions). Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: 6 months
Population: One participant not analyzed as they never received study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Colorectal Cancers Metastasized to the Liver
Number analyzed (Participants) | 13
Months | NA [NA to NA] — No participants progressed in 6 months.

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, an average of 28 months and 23 days.
Population: One participant never received study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Cancers Metastasized to the Liver
Number analyzed (Participants) | 13
Participants | 13

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, an average of 28 months and 23 days.
Arm/Group | Colorectal Cancers Metastasized to the Liver
All-Cause Mortality (participants affected / at risk) | 12/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colorectal Cancers Metastasized to the Liver (N=14)
Blood and lymphatic system disorders - Other, Spleen infarction (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Pain (General disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colorectal Cancers Metastasized to the Liver (N=14)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Activated partial thromboplastin time prolonged (Investigations) | 8 (14)
Alanine aminotransferase increased (Investigations) | 3 (4)
Alkaline phosphatase increased (Investigations) | 7 (10)
Anemia (Blood and lymphatic system disorders) | 8 (21)
Anorexia (Metabolism and nutrition disorders) | 5 (6)
Anxiety (Psychiatric disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 6 (9)
Chills (General disorders) | 4 (5)
Confusion (Psychiatric disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Edema limbs (General disorders) | 3 (3)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Fatigue (General disorders) | 11 (16)
Fecal incontinence (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 5 (14)
Flu like symptoms (General disorders) | 6 (9)
Headache (Nervous system disorders) | 4 (4)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (10)
Hypokalemia (Metabolism and nutrition disorders) | 6 (10)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3)
Lymphocyte count decreased (Investigations) | 7 (17)
Lymphocyte count increased (Investigations) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Soreness in shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (11)
Neck edema (General disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 5 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 6 (13)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Dermatitis/Erythematous rash on bilateral shins with dry skin
Skin and subcutaneous tissue disorders - Other, Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (12)
Weight loss (Investigations) | 2 (4)
White blood cell decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT04166383/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT04166383/ICF_001.pdf